CLINICAL TRIAL: NCT05609318
Title: Study of Tissue Iron Uptake in Iron-Deficient Patients Receiving Intravenous Iron Replacement Therapy: A Prospective Observational Study (STUDY)
Brief Title: Imaging Intravenous Iron
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: PID16038
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-11

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- iron-deficient: patients prescribed intravenous iron infusion for the treatment of iron deficiency as part of standard clinical care

SUMMARY:
The aim of this study is to track where the iron goes in different tissues in the hours, days and weeks after an intravenous iron infusion. We will track iron in tissues using MRI relaxometry parameters R1/R2/R2* which are well established as accurate indicators of tissue iron content.

DETAILED DESCRIPTION:
This is a prospective, observational, study exploring the kinetics of tissue iron uptake following intravenous iron infusion (Ferinject), received as part of standard clinical care in a group of iron-deficient patients.

Participants will be recruited through the Iron Deficiency Management Service, part of the Oxford University Hospitals NHS Foundation Trust (OUHFT) . Participants will receive their intravenous iron infusion (Ferinject) as part of their standard clinical care by an NHS clinician. They will undergo all the study MRI scans and additional study procedures at the Oxford Centre for Clinical Magnetic Resonance Research (OCMR), which is based at the John Radcliffe Hospital and is part of the Division of Cardiovascular Medicine within the Radcliffe Department of Medicine at the University of Oxford.

Each participant will undergo 4 MRI scans; baseline, 3hours, 14 days and 42 days post intravenous iron infusion. Blood samples will also be collected at those timepoints for assessment of relevant heamatological and iron parameters.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Aged 18 years or above.
* Anaemia (haemoglobin less than 120g/L for women and less than 130g/L for men) and/or confirmed iron deficiency (ferritin less than 100mcg/L and/or transferrin saturation less than 20%).
* Scheduled to receive intravenous iron for correction of iron deficiency.

Exclusion Criteria:

* Any MRI incompatible implants (e.g. cardiac, neuro, ocular implants, surgical clips, aneurysm clips, shrapnel/bullets)
* Pregnant or lactating participant
* Acute decompensated heart failure
* Unstable clinical status
* Any other medical conditions which would influence the reliability of the study results determined by the investigators.
* Any other contraindication to MRI to be confirmed by the qualified MRI operator, e.g. tattoos containing traces of metal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are patients who require intravenous iron as part of their standard clinical care. They will be recruited from referrals to the Iron Deficiency Management Service (IDMS), part of Oxford University Hospitals NHS Foundation Trust (OUHFT). This service receives referrals from multiple sources across Oxfordshire.
  Patient referrals will be screened by members of the NHS Clinical team at IDMS to identify potentially eligible participants.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-10-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To establish the kinetics of iron uptake into the heart, liver, spleen, kidney, skeletal muscle and blood following a single intravenous iron infusion (Ferric carboxymaltose, Ferinject, 1000mg) | baseline, 3hr, 14 days and 42 days post intravenous iron infusion
  Changes from baseline in multi-organ magnetic resonance relaxometries (delta R1/R2/R2* (seconds) for each participant.

SECONDARY OUTCOMES:
Determine the effects of iron infusion (Ferric carboxymaltose, Ferinject, 1000mg) on serum iron indices and serum markers of tissue iron damage. | baseline, 3hr, 14 days and 42 days post intravenous iron infusion
  Change from baseline in:
  1. Serum iron indices: iron (uM), ferritin (mg/L), transferrin saturation (%), non-transferrin bound iron (uM)
  2. Serum markers of tissue iron damage, including but not limited to lipid peroxidation markers malondialdehyde (MDA in mM) and 4-Hydroxynonenal (HNE in mM)

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Centre for Clinical Magnetic Resonance Research (OCMR), Oxford, Oxfordshire, United Kingdom